CLINICAL TRIAL: NCT03114709
Title: Mindful Movement for Physical Activity and Wellbeing in Older Adults: A Community Based Randomized Hybrid Effectiveness-Implementation Study
Brief Title: Mindful Movement for Physical Activity and Wellbeing in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: YMCA (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 1611S99323-2; R21AT009110 (NIH)
Record Dates: First submitted 2017-03-07; First posted 2017-04-14 (Actual); Last update posted 2019-11-01 (Actual); Status verified 2019-10

CONDITIONS: Physical Inactivity
Keywords: Mindfulness; Exercise; Physical activity; Behavior change; Aging; Randomized controlled trial; Pilot
MeSH Terms: conditions — Sedentary Behavior; Motor Activity | interventions — Health

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindful Movement (Experimental): 8, 90-minute, in-person, group sessions over 8 weeks
  Interventions: Other: Mindful Movement
- 10 Keys to Health & Wellbeing (Active Comparator): 8, 90-minute, in-person, group sessions over 8 weeks
  Interventions: Other: 10 Keys to Health & Wellbeing

INTERVENTIONS:
Other: Mindful Movement — The program focuses on enhancing individuals' mindfulness capabilities and skills, specifically attention regulation, body awareness, emotional regulation, and shifts in self-perception, by providing opportunities for education, practice, and social support in mindfulness practices and physical activity.
  Arms: Mindful Movement
Other: 10 Keys to Health & Wellbeing — This community-based educational program provides participants useful content focused on general health related topics including common chronic conditions, social support, social participation, cancer screening, immunization and keeping active.
  Arms: 10 Keys to Health & Wellbeing

SUMMARY:
Physical inactivity has reached pandemic proportions and is associated with increased morbidity, mortality, and healthcare costs. Of particular concern is that most middle to older age adults fall far short of recommendations for health enhancing physical activities. This research takes a novel approach to tackling this problem by combining mindfulness with behavioral strategies in a unique 'Mindful Movement' program offered through YMCA community facilities.

DETAILED DESCRIPTION:
Physical inactivity in the United States has become a critical public health concern for all age groups. With a large segment of the population rapidly aging, there is growing interest in ensuring mid to older age adults (50+) stay active and reduce sedentariness, to decrease their morbidity and mortality risk. While older adults are advised to engage in at least 150 minutes/week of moderate to vigorous physical activity (PA), most do not. Specific theory based behavioral strategies have been shown to positively affect health and activity behaviors. There is also emerging evidence that mindfulness based interventions (MBI) may facilitate PA through increased mind-body awareness and self-regulation. However, research for MBIs and physical activity is currently limited, both in quantity and methodological rigor.

The broad long-term objective is to optimize physical and sedentary activity levels in middle-older age adults through an integrated mindfulness and behavioral approach scalable for broad dissemination. The University of Minnesota (UMN) will work with the YMCA Greater Twin Cities, a community based organization committed to providing accessible resources to "build healthy spirit, mind and body for all" and making healthy aging a priority. To decrease time between discovery and translation, a two-phase hybrid effectiveness-implementation design will be used.

Phase I will address the following: 1) project organization, barrier/facilitator assessment, protocol development, and training; and 2) evaluation of feasibility of project protocols at multiple levels in a randomized pilot study (n=30) of Mindful Movement versus a modified 10 Keys to Health & Wellbeing educational control using transition milestones.

Phase II will address: 1) investigation of the relative effectiveness of Mindful Movement versus control in a full-scale randomized controlled trial (RCT, n=182) using accelerometer based PA at 9 weeks (primary outcome) and at 26 and 52 weeks (secondary outcomes) as well as other secondary measures include sedentary activity, quality of life, exercise self-efficacy and expectations, mindfulness, wellbeing, bodily pain, and adverse events; and 2) RCT interpretation by providing contextual data from participants, staff, and organizational leadership. These will include: enrollment, adherence, follow up, and fidelity rates; and perceptions of barriers/facilitators, relevance, practicality, affordability and acceptability. This information will be used to create a toolkit for implementation at other YMCA sites.

This project is innovative in that it will be among the first to assess MBIs for enhancing older adults' physical activity in community based settings using a design intended to facilitate and accelerate research translation. Through the UMN and YMCA partnership, there is great potential to develop a sustainable and replicable physical activity intervention with meaningful impact and nationwide reach.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 50 years of age
* Accelerometer wear time ≥10 hours on at least 4 days in a 7 consecutive day period between baselines
* Self-report of <140 minutes of MVPA per week in 3 months prior to baseline AND accelerometer recorded <100 minutes of MVPA between baselines
* Mini-Mental State score ≥ 24
* Independent self-ambulation
* Provides consent and is willing to participate in data collection activities

Exclusion Criteria:

* Pregnancy
* Unwilling or unable to participate in study activities
* Current or upcoming participation in educational programs similar to those under study
* Medical restrictions to increasing Moderate Vigorous Physical Activity (MVPA) AND health care provider does not provide clearance
* Terminal illness
* Contraindications to mindfulness practice

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-03-27 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2019-02-28 (Actual)

PRIMARY OUTCOMES:
Moderate-Vigorous Physical Activity (MVPA) | Change score: 9 weeks score - baseline score
  Minutes/week spent in ≥10-min bouts of MVPA

SECONDARY OUTCOMES:
Quality of Life-Euroqol 5D (EQ5D) | 0, 9 weeks
  The EQ5D captures five dimensions of health (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) over 5 levels (no problem, slight problem, moderate problem, severe problem, unable to perform/extreme problem).
Exercise Self-Efficacy- Self-Efficacy for Exercise (SEE) scale | 0, 9 weeks
  Individuals are asked to rate their confidence in their ability to exercise. Confidence ratings range from 0 (not confident) to 10 (very confident).
Exercise Expectations-Outcome Expectations for Exercise-2 (OEE-2) scale | 0, 9 weeks
  This is a 13-item instrument focused on beliefs about the positive and negative physical and mental health benefits of exercise. Responses range from 1 (strongly agree) to 5 (strongly disagree).
Mindfulness- Mindful Attention Awareness Scale (MAAS), Frieberg Mindfulness Inventory (FMI) | 0, 9 weeks
  The MAAS scale is comprised of 15 items measured on a 6-point scale (1=almost always, 6=almost never). The FMI addresses 14 items with a four-point response scale (1=rarely, 4=almost always).
Wellbeing-8-item Flourishing Scale | 0, 9 weeks
  This scale assesses perceived success in relationships, self-esteem, and purpose.
Pain-11 box numerical rating scale | 0, 9 weeks
  An 11-box numerical rating scale (0=no pain, 10=the worst pain possible) will be used for spinal pain, and upper and lower extremities.
Social Connectedness & Assurance | 0, 9 weeks
  This includes two, eight-item questionnaires with a six-item scale (strongly agree, strongly disagree).
Physical Activity-International Physical Activity Questionnaire (IPAQ) | 0, 9 weeks
  An adapted, nine-item instrument addressing days/week and minutes/day spent on physical activity in the past 7 days is used to measure physical activity.
Satisfaction | 9 weeks
  Participants will rate their overall satisfaction (satisfied, completely dissatisfied) with the intervention.
Intervention Barriers | Planning phase, 0, 9 weeks
  This qualitative, open ended assessment explores barriers to participation in the intervention.
Intervention Facilitators | Planning phase, 0, 9 weeks
  This qualitative, open ended assessment explores facilitators to participation in the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Roni Evans, PhD, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - YMCA Southdale, Edina, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - YMCA Midway, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Data will be provided in aggregate.